CLINICAL TRIAL: NCT05415579
Title: Demyelinating Diseases of the Central Nervous System Registry for Patients With Traditional Chinese Medicine (DATE-TCM)
Status: Not yet recruiting | Type: Observational
Sponsor: Dongzhimen Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Ying Gao, Professor, Dongzhimen Hospital, Beijing
Other Study IDs: DDCR-TCM-2022
Record Dates: First submitted 2022-06-09; First posted 2022-06-13 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Demyelinating Diseases of the Central Nervous System (DDC)
Keywords: Demyelinating Diseases of the Central Nervous System; Multiple sclerosis; Neuromyelitis optica spectrum disorder; Myelin oligodendrocyte glycoprotein associated disorder
MeSH Terms: conditions — Demyelinating Diseases; Multiple Sclerosis; Neuromyelitis Optica | interventions — Medicine, Chinese Traditional

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- DDC patients with Traditional Chinese medicine (TCM) treatment: TCM treatment includes Chinese herbal medicine, acupuncture, moxibustion, massage, taiji, and qigong.
  This study does not limit Western medical treatment methods. Patients commonly applied high dose of intravenous steroid treatment in the acute phase, which usually referred to intravenous administration of 1g or 500mg of glucocorticoid daily for 3 consecutive days and reduced by half every 3 days. In addition, plasma exchange and immunoabsorption are also optional treatment for the acute phase. Immunomodulatory therapies including low dose of steroid, immunosuppressants (Azathioprine, Mycophenolate, etc.), and disease-modifying therapy (fingolimod, Teriflunomide, Rituximab, Satralizumab, etc.) are necessary for the remission phase.
  Interventions: Other: Traditional Chinese medicine (TCM)

INTERVENTIONS:
Other: Traditional Chinese medicine (TCM) — TCM treatment includes Chinese herbal medicine, acupuncture, moxibustion, massage, taiji, and qigong.

SUMMARY:
Demyelinating Diseases of the Central Nervous System Registry for Patients with Traditional Chinese Medicine (DATE-TCM) is an observational study aiming to better define the multidimensional (epidemiologic, demographic and clinical) characteristics of Demyelinating Diseases of the Central Nervous System (DDC) patients receiving Traditional Chinese medicine (TCM) treatment, the type and long-term safety and effectiveness of TCM in DDC populations, as well as the interaction of TCM treatment and disease-modifying therapy in the management of DDC.

DETAILED DESCRIPTION:
Demyelinating Diseases of the Central Nervous System (DDC) is a collective term for a group of immune-mediated disorders including multiple sclerosis, Neuromyelitis optica spectrum disorder, and myelin oligodendrocyte glycoprotein associated disorder, characterized by myelin loss and axonal damage in the central nervous system. Traditional Chinese medicine (TCM), a main form of complementary and alternative medicine provides a potential possibility to DDC management and has been applied to a considerable number of patients with this disorder in China as well as in other regions or countries worldwide. Demyelinating Diseases of the Central Nervous System Registry for Patients with Traditional Chinese Medicine (DATE-TCM) provides a prospective and voluntary registry aiming to include 2000 eligible adult DDC patients with TCM intervenes from around 30 participating centers by using a web-based system. Baseline data will be recorded and subsequently regular follow-up visits will be implemented every 3-6 months for a total of 5 years. Main objective of DATE-TCM is to create an organized multicenter structure to collect reliable data for better define the multidimensional (epidemiologic, demographic and clinical) characteristics of DDC patients receiving TCM treatment, the type and long-term safety and effectiveness of TCM in DDC populations, as well as the interaction of TCM treatment and disease-modifying therapy in the management of DDC.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants with aged 18-65 years old; Diagnosis of DDC including multiple sclerosis (MS), Neuromyelitis optica spectrum disorder (NMOSD), and myelin oligodendrocyte glycoprotein-associated disease(MOGAD) according to relevant criteria or consensus; Patients who receive or are willing to receive TCM treatment including the Chinese herbal medicine, acupuncture, moxibustion, massage, taiji, and qigong; Informed written consent obtained from the patient, and/or his/her legally authorized representatives.

Exclusion Criteria:

* Refusal to give informed consent; Malignancies, infectious diseases (HBV, HCV, HIV, etc.), congenital or acquired severe immunodeficiency, significant cardiovascular, pulmonary, and hepatic diseases or conditions; Mental disturbance or severe cognitive impairment impeding necessary information gathering and assessment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: DATE-TCM includes all patients with Demyelinating Diseases of the Central Nervous System at beginning of study.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-06-20 (Estimated); Primary Completion 2029-10-31 (Estimated); Study Completion 2030-05-31 (Estimated)

PRIMARY OUTCOMES:
Annualized Aggregate Relapse Rate (ARR) | Baseline up to 5 years
  ARR is defined as the number of confirmed relapses in a year. A relapse is defined as the appearance of a new or worsening of a previously stable or improving pre-existing neurological abnormality, separated by at least 30 days from onset of a preceding relapse. The abnormality must be present for at least 24 hours and occur in the absence of fever or infection. The ARR was the mean of the annualized ARRs for all patients, calculated as the total number of confirmed relapses divided by the total number of days on study multiplied by 365.25.

SECONDARY OUTCOMES:
Total Number of Adverse Events During Evaluation | Baseline up to 5 years
  Adverse Events (AE) are any unfavorable and unintended sign, symptom, syndrome, or illness observed by the investigator or reported by the participant during the study.
Percentage of Participants With Adverse Events | Baseline up to 5 years
  Adverse Events (AE) are any unfavorable and unintended sign, symptom, syndrome, or illness observed by the investigator or reported by the participant during the study.
Time to 3-month Sustained Disability Progression | 5 years
  3-month sustained disability progression (DP) was defined as an increase from baseline of at least 1-point in EDSS score (at least 0.5-point for participants with baseline EDSS score >5.5) that persisted for at least 3 months.
  EDSS scale ranges from 0 (Normal neurological exam, no disability) to 10 (Death) in 0.5 unit increments that represent higher levels of disability. Scoring is based on an examination by a neurologist. Kaplan-Meier method consists in computing probabilities of non-occurrence of event at any observed time of event and multiplying successive probabilities for time ≤t by any earlier computed probabilities to estimate the probability of being event-free for the amount of time.
Time to 6-month Sustained Disability Progression | 5 years
  6-month sustained disability progression (DP) was defined as an increase from baseline of at least 1-point in EDSS score (at least 0.5-point for participants with baseline EDSS score >5.5) that persisted for at least 6 months.
  EDSS scale ranges from 0 (Normal neurological exam, no disability) to 10 (Death) in 0.5 unit increments that represent higher levels of disability. Scoring is based on an examination by a neurologist. Kaplan-Meier method consists in computing probabilities of non-occurrence of event at any observed time of event and multiplying successive probabilities for time ≤t by any earlier computed probabilities to estimate the probability of being event-free for the amount of time.
Number of New or Newly Enlarging T2 hyperintense lesions as Measured by Magnetic Resonance Imaging (MRI) | From baseline to 12 months, 24 months, 36 months, 48 months, 60 months
  The number of new or newly enlarging T2 hyperintense lesions that developed in each subject compared to baseline assessed on magnetic resonance imaging (MRI) scans. The estimates of mean T2 hyperintense lesion count were calculated from a negative binomial regression model adjusted for region and baseline T2 hyperintense lesion volume.
Number of Gadolinium-enhancing T1-weighted Lesions as Measured by Magnetic Resonance Imaging (MRI) | From baseline to 12 months, 24 months, 36 months, 48 months, 60 months
  The number of Gd-enhancing lesions was assessed by using MRI scans following administration of gadolinium, a contrast agent.
Percent Change in Brain Volume Measured by Magnetic Resonance Imaging (MRI) | From baseline to 12 months, 24 months, 36 months, 48 months, 60 months
  Calculations of brain volume change were performed using the structural image evaluation of normalized atrophy (SIENA), software included in the Functional Magnetic Resonance Imaging of the Brain (FMRIB) software library.
Change in Multiple Sclerosis Functional Composite (MSFC) score | Every 6 months up to 5 years
  The Multiple Sclerosis Functional Composite (MSFC) is a multidimensional clinical outcome measure that includes quantitative tests of leg function/ambulation (Timed 25-Foot Walk), arm function (9-Hole Peg Test), and cognitive function (Paced Auditory Serial Addition Test).
Change in Symbol Digit Modalities Test (SDMT) score | Every 6 months up to 5 years
  The SDMT measures the time to pair abstract symbols with specific numbers. The test requires elements of attention, visuoperceptual processing, working memory, and psychomotor speed. The score is the number of correctly coded items from 0-110 in 90 seconds. The total score provides a measure of the speed and accuracy of symbol-digit substitution.
Chance in fatigue severity scale (FSS) score | Every 6 months up to 5 years
  FSS is a short questionnaire that requires patient to rate level of fatigue.
Change in EuroQol- 5 Dimension (EQ-5D) score | Every 6 months up to 5 years
  The EQ-5D descriptive system is a preference-based HRQL measure with one question for each of the five dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. A mixed effect model for repeated measures was used for this analysis. An unstructured covariance was used to model within-participant error.
Change from Multiple Sclerosis impact scale (MSIS) score | Every 6 months up to 5 years
  The MSIS-29 is a disease specific patient-reported outcome measure that has been developed and validated to examine the physical and psychological impact of MS from a patient's perspective; it measures 20 physical items and 9 psychological items. A mixed effect model for repeated measures was used for this analysis. An unstructured covariance was used to model within-participant error.